CLINICAL TRIAL: NCT06903923
Title: Bone Metabolism in Adolescents Undergoing GLP-1 Receptor Agonist Therapy
Brief Title: Bone Metabolism in 12-21 Year Olds Undergoing GLP-1 Receptor Agonist Therapy
Status: Recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Madhusmita Misra, Professor of Pediatrics, University of Virginia
Other Study IDs: HSR302394; R01HD118635 (NIH)
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-03

CONDITIONS: Obesity in Children; Bone Strength; GLP - 1; Lifestyle Modification; Bone Density; Obesity
Keywords: obesity; obesity in children; bone strength; GLP-1; Lifestyle modification; bone density; semaglutide
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- GLP-1 receptor agonist (RA)/semaglutide + Calcium & Vitamin D: The GLP-1 RA, semaglutide, will be prescribed by the participants' physician for routine clinical care for the management of obesity while the Calcium + Vitamin D will be provided by the research investigator.
  Interventions: Drug: GLP-1 receptor agonist
- Lifestyle Management + Calcium & Vitamin D: The Lifestyle Management will be overseen by the participants' physician for routine clinical care for the management of obesity while Calcium + Vitamin D will be provided by the research investigator.
  Interventions: Behavioral: Lifestyle Management

INTERVENTIONS:
Drug: GLP-1 receptor agonist — Participants prescribed a GLP-1 receptor agonist (semaglutide) by their physician will be enrolled in this arm of the study. All participants will receive study provided calcium & vitamin D supplement to support bone health and to reduce this as a confounding factor in overall outcomes
  Groups: GLP-1 receptor agonist (RA)/semaglutide + Calcium & Vitamin D
Behavioral: Lifestyle Management — Participants receiving usual lifestyle interventions will be enrolled in this arm of the study. All participants will receive study provided calcium & vitamin D supplement to support bone health and to reduce this as a confounding factor in overall outcomes
  Groups: Lifestyle Management + Calcium & Vitamin D

SUMMARY:
The goal of this clinical trial is to compare bone health markers over 24 months in participants 12 - 21 years of age with obesity who are starting the glucagon-like peptide-1 (GLP-1) Semaglutide as compared to those with similar weight followed by lifestyle management.

Participants will:

* Take Semaglutide as prescribed or continue to work on lifestyle management for weight loss
* Take provided calcium and vitamin D supplements
* Attend 6 study visits over 24 months with two at the beginning and then every 6 months that include:

  * History and Physical Exams
  * Lab Work
  * Imaging studies
  * Questionnaires
  * 24-hour dietary recalls
  * Mixed Meal Tolerance Test with a nutritional energy drink and six blood draws

DETAILED DESCRIPTION:
Obesity is now epidemic, and as a consequence, the use of weight loss medications and surgery to manage obesity is increasing. Weight loss surgery is associated with significant bone loss, concerning during the adolescent years of peak bone accrual. With the increasing use of weight loss medications, particularly glucagon-like-peptide 1 receptor agonists (GLP-1 RAs), in adolescents, it is essential to determine whether weight loss following use of these medications is associated with detrimental effects on skeletal health. Data from the literature are conflicting following use of semaglutide (a commonly used GLP-1 RA) in adults with obesity. Whether GLP-1 RA use preserves bone anabolic activity during adolescence merits investigation and is the focus of the proposal. If the investigators' hypotheses prove correct and use of GLP-1 RAs preserves bone accrual and skeletal health in youth with obesity, the results of this study may favor GLP-1 RA treatment over surgery following lifestyle management. Multiple mechanisms contribute to bone loss after surgery in youth including mechanical unloading of bone from weight loss, loss of lean mass, and changes in hormones that stimulate anabolic bone activity and/or are anti-resorptive. Weight loss following use of GLP1-RAs should similarly lead to skeletal unloading, reductions in lean mass, and changes in hormones. However, GLP-1 RAs have direct bone anabolic effects, and anti-resorptive effects as demonstrated in both rodent and human studies. Thus, GLP-1 RAs might mitigate deleterious effects of weight loss on skeletal health through a direct impact on bone formation and resorption. DXA-based BMD measurements have limitations in obesity and during weight loss, being susceptible to artifactual changes from a reduction in soft tissue thickness after severe weight loss. The study will therefore use advanced 3D imaging techniques to overcome limitations of DXA in the context of the marked soft tissue changes following weight loss. The investigators' overall hypothesis is that despite marked weight loss in adolescents with obesity receiving GLP-1 RAs (specifically semaglutide, an FDA approved, commonly used GLP-1 RA in youth) over 24 months, study participants will demonstrate preservation of areal and volumetric BMD, bone geometry, structure and estimated strength, and improvements in estimated fracture risk.

Aim 1: To determine to what extent GLP-1 RA therapy alters bone density, geometry, structure, strength and load-to-strength ratio prospectively over 24 months in adolescents and young adults ages 12-21 years with obesity compared to controls of similar weight followed with lifestyle management. The investigators hypothesize that following GLP-1 RA (semaglutide) therapy vs. lifestyle management:

Hypothesis 1A: Volumetric BMD of the distal radius (a non-weight bearing site) (primary endpoint) and distal tibia (a weight-bearing site) by HRpQCT, and areal BMD of the hip and spine by DXA will be preserved.

Hypothesis 1B: Cortical and trabecular geometry and structure at the distal radius and tibia (by HR-pQCT), and bone strength estimates (by μFEA) will be preserved; load-to-strength ratio will improve.

Aim 2: To investigate novel physiologic mechanisms mediating maintenance of skeletal integrity following use of semaglutide.

Hypothesis 2: The investigators hypothesize that preservation of skeletal health despite reductions in weight, lean mass, ghrelin, insulin, oxytocin and estrone and increases in sclerostin is associated with increases in bone formation (as assessed by P1NP, a marker of bone formation) that equal or exceed those of bone resorption (as assessed by CTX, a marker of bone resorption), indicative of balanced bone turnover and net skeletal stability.

Adolescence is a critical time for bone accrual and the use of both GLP-1 RAs and MBS is increasing in youth. The study will provide novel data needed to establish whether use of GLP-1 RAs prevents the impairment in skeletal health observed following surgery in youth. Clarifying these mechanisms will identify optimal weight loss strategies in youth with obesity following lifestyle intervention.

Design: This is a non-randomized two-group parallel observational pragmatic trial. The study will recruit 120 adolescents and young adults with obesity 12-21 years old, 60 of whom are being started clinically on semaglutide therapy and 60 who will be followed with 'usual' care. Participants will be matched for BMI, sex, self-described race, age, and pubertal stage. Normally menstruating females will be studied during the first 10 days of their cycles. The baseline visit will occur before starting semaglutide therapy (for the active arm), and will be followed by visits 6, 12, 18, and 24-months after starting therapy. Controls will be followed at the same frequency. Participants will be counseled regarding lifestyle measures per protocol ('usual' care).

Analytical Plan:

Data generated will be longitudinal over 12 and 24-months. There are two study groups for the longitudinal component: those undergoing semaglutide therapy, and adolescents with obesity followed with usual care.

Analysis of Treatment Group Comparability: Demographic and baseline characteristics will be summarized by treatment group (semaglutide vs. usual care) using descriptive statistics and will be compared using a t-test or Chi-square test depending on data types.

Analysis of Aim 1:

The study is powered for analysis of the primary endpoint i.e. baseline to 24-month change in the HR-pQCT measure of total vBMD (distal radius). This analysis will include all randomized subjects according to treatment (intent to treat). The investigators will test for equivalency of the between-group treatment effects by examining if the upper limit of the 90% confidence interval of the semaglutide versus 'usual care' difference in the group-specific HR-pQCT mean change is above -30 (i.e., no less than 10% below 300 mgHA/cm3) and the lower limit is below 30 (i.e., no more than 10% above 300 mgHA/cm3). The same analysis approach as that of the primary endpoint analysis will be applied to secondary endpoints. Investigators will not adjust Type-1 error for the inference of these multiple secondary endpoints.

Method to analyze longitudinal data: Although the primary analysis endpoints are 24-month change, for longitudinal data collected at multiple time points (baseline, 12 and 24 months), as parallel analyses, investigators will utilize all available repeated measures in longitudinal general linear mixed effects models with the treatment difference at 24-month as the primary contrast of interest. The subject level intercept will be considered as random. The closest pattern of time dependency will be identified by means of exploratory longitudinal plots before fitting the model. The model will include group and time as the main effects and group x time as the interaction, and the above-mentioned equivalency test method will be applied to the model-based estimate of the treatment difference at 24-month. SAS Proc Mixed procedure with exchangeable- or more appropriate correlation structure will be used. This analysis will include all data collected on all subjects irrespective of whether the subject completed all 24 months of follow up, and follows the Institute of Medicine (IOM) suggestion for analysis of data with missing observations. We will adjust for confounders as necessary (the study will match participants for age, sex, race, and BMI). For Aim 2, the investigators will estimate within-group correlations (Pearson or Spearman as appropriate based on distribution) of 24-month change in weight, lean mass, and hormones with change in P1NP and CTX; and then examine if these correlations differ between the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults 12 - 21 years old starting semaglutide therapy or followed by usual care/lifestyle management
* Diagnosis of obesity (BMI ≥ 95th percentile for age and sex)
* Participants on semaglutide must have demonstrated efforts at weight loss with "usual care," and consistent compliance with appointments and recommendations.
* Participants must demonstrate sufficient maturity, psychological stability and cognitive capacity to recognize the significance of being on medical therapy and implement required behavioral changes.

Exclusion Criteria:

* Current or previous history of pregnancy and breast feeding
* Personal or family history of medullary thyroid cancer or multiple endocrine neoplasia type 2 if in the GLP-1 RA group
* Less than 5 kg weight change over 3 months given the known impact of significant weight loss on bone density
* Use of medications such as metformin, phentermine, or topiramate that may cause weight loss, or antipsychotic medications that may cause weight gain if treated for <6 months, or if dosage is not stable for >2 months
* Medications other than calcium or vitamin D that affect bone, such as glucocorticoids, phenytoin, phenobarbitone (unless there is a washout period of 3 months prior to enrollment if discontinuation is medically permissible); female participants on hormonal contraception will be excluded if this involves use of depot medroxyprogesterone acetate (given its profound deleterious effect on bone density); however, those on combined oral contraceptives, continuous oral progestin, a progestin releasing intrauterine device or implant will not be excluded
* Untreated thyroid dysfunction or on stable dose for <3 months
* Medical conditions known to impact weight or bone density, such as chronic gastrointestinal disorders (including inflammatory bowel disease), other inflammatory conditions, such as rheumatoid arthritis or ankylosing spondylitis, untreated thyroid disease, and hypercortisolemia
* HbA1C >8% (to avoid deleterious effects on bone from uncontrolled T2DM)
* Smoking >10 cigarettes/day given deleterious effects on bone; substance abuse per DSM-5
* Weight >450 lbs due to limits for DXA scanners
* Judged by the investigators to be inappropriate for the study for other reasons not detailed above.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, teenagers and adults with obesity 12-21 years old
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in total volumetric bone mineral density (vBMD) the distal radius measured by HR-pQCT | 24 months
  To assess the effect of GLP-1 RA (semaglutide) therapy on vBMD at a non-weight-bearing site (distal radius) in adolescents and young adults with obesity, compared to matched controls receiving lifestyle management.

SECONDARY OUTCOMES:
Change in total volumetric bone mineral density (vBMD) the distal tibia measured by HR-pQCT | 24 months
Change in trabecular vBMD of the distal tibia and radius assessed by HR-pQCT | 24 months
Change in areal BMD of the lumbar spine and total hip measured by DXA | 24 months
Change in estimated bone strength (radius and tibia) using micro finite element analysis (μFEA) | 24 months
Change in load-to-strength ratio at the radius and hip | 24 months
Change in bone turnover markers (P1NP and CTX) | 24 months
  To assess whether preservation of skeletal integrity is associated with changes in bone formation and resorption markers (P1NP and CTX), and to explore potential mediating mechanisms such as changes in weight, lean mass, ghrelin, insulin, oxytocin, estrone, and sclerostin.
Changes in gut related and sex hormones | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Madhusmita Misra, MD, MPH, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Medical Center, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Primary and secondary endpoint data, including all bone endpoints, will be submitted to the Harvard Dataverse repository to enable other researchers to analyze our study data independently. The privacy, rights, and confidentiality of human research participants will be protected by sharing only de-identified data.
Supporting Information: SAP, ICF
Time Frame: Data sharing will occur no later than the end of performance period of the extramural award that generated the data. There is no end date planned at this time.
Access Criteria: Study investigators will make access to deidentified data available via repository without restriction to access. Data available will include deidentified demographic data and those related to primary and secondary endpoints.